CLINICAL TRIAL: NCT03955315
Title: A Randomized, Double Blind, Sham-controlled, Multi-center Phase I / II Clinical Study to Assess the Safety and Efficacy of IDCT in Patients With Lumbar Degenerative Disc Disease
Brief Title: Study to Evaluate the Safety and Preliminary Efficacy of IDCT, a Treatment for Symptomatic Lumbar Disc Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DiscGenics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DGX-J01
Record Dates: First submitted 2019-05-14; First posted 2019-05-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2022-11

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High Dose IDCT (Experimental): Single intradiscal injection with High Dose IDCT (9M cells)
  Interventions: Biological: IDCT
- Low Dose IDCT (Experimental): Single intradiscal injection with Low Dose IDCT (3M cells).
  Interventions: Biological: IDCT
- Sham (Sham Comparator): Sham needle puncture (outside disc)
  Interventions: Procedure: Sham

INTERVENTIONS:
Biological: IDCT — Discogenic Cells + Sodium Hyaluronate Vehicle
  Other Names: Injectable Disc Cell Therapy
  Arms: High Dose IDCT; Low Dose IDCT
Procedure: Sham — Needle puncture under the muscular layer in front of the intervertebral disc
  Arms: Sham

SUMMARY:
The purpose of this study is to compare the safety and preliminary efficacy of intradiscal injections of two doses of IDCT (Discogenic Cells + Sodium Hyaluronate vehicle) and one sham control in subjects with chronic low back pain due to Degenerative Disc Disease (DDD) at one lumbar level from L3 to S1.

DETAILED DESCRIPTION:
This is a Phase I, randomized, double-blind, sham-controlled, parallel-group, multi-center study in subjects with single-level, symptomatic lumbar intervertebral disc degeneration (>6 months) and unresponsive to conservative therapy for at least 3 months. The study will compare single intradiscal injections of high and low dose IDCT with one sham control group.

6 study visits will be completed by all subjects; screening, day 1 (injection day), week 4, week 12, week 26 and week 52. The subject will be assessed for safety and efficacy utilizing VAS, ODI and JOABPEQ questionnaires alongside radiographic evaluations. The study will have a 6 month follow-up and a 6 month extension period (total 1 year).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of early to moderate degenerative disc disease (DDD), Modified Pfirrmann Grade 3-7.
* Chronic low-back pain for at least 6 months prior to screening; unresponsive to at least 3 months of conservative care.
* Low-back pain of 40 to 90 mm on the VAS
* ODI score of 30 to 90.

Exclusion Criteria:

* Symptomatic involvement of more than one lumbar disc.
* Other persistent pain/nerve issues including, for example, radiculopathy, leg pain, Cauda Equine syndrome, etc.
* Fracture of the spine, previous lumbar spine surgery or previous treatment of the target disc.
* Evidence of dynamic instability on lumbar flexion-extension radiographs.
* Grade 2 or higher spondylolisthesis at the target disc, lumbar spondylitis or other undifferentiated spondyloarthropathy, or Type III Modic changes around the target disc.
* Clinical suspicion of a full thickness annular tear at the target disc or other abnormal disc morphology.
* Subjects who test positive for communicable disease, have significant systemic disease, or are prone to infection.
* Patients who are deemed unsuitable for clinical study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Safety as measured by number of Adverse Events | 1 year
  To evaluate the safety and tolerability of a single injection of IDCT in subjects with single-level, symptomatic early to moderate lumbar intervertebral disc degeneration as measured by the incidence of AEs and SAEs observed from Day 1 to week 52
Efficacy (Pain): Visual Analogue Scale (VAS) | 6 months
  Evaluate the effect of IDCT on pain as measured by a 0-100mm Visual Analogue Scale (VAS). 0: no pain, 100: worst pain imaginable

SECONDARY OUTCOMES:
Disability | 1 year
  Evaluate the effect of IDCT on disability as measured by the Oswestry Disability Index (ODI). Score of 0%: no disability, score of 100%: severely disabled
Efficacy (Pain): JOABPEQ | 1 year
  Evaluate the effect of IDCT on pain as measured by JOABPEQ. The range of the score for each domain is from 0 to 100, with higher scores indicating a better condition.

OTHER OUTCOMES:
Radiographic Assessments | 1 year
  To evaluate morphologic changes of treated intervertebral discs using MRI & X-Ray assessments.

CONTACTS AND LOCATIONS:
Locations (6):
- Japan (6):
  - Chiba University Hospital, Chuo-ku, Chiba
  - Tokai University Hospital, Isehara, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - Nagoya university hospital, Shōwaku, Nagoya
  - Osaka University Hospital, Suita, Osaka
  - University of Yamanashi Hospital, Chūō, Yamanashi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silverman LI, Dulatova G, Tandeski T, Erickson IE, Lundell B, Toplon D, Wolff T, Howard A, Chintalacharuvu S, Foley KT. In vitro and in vivo evaluation of discogenic cells, an investigational cell therapy for disc degeneration. Spine J. 2020 Jan;20(1):138-149. doi: 10.1016/j.spinee.2019.08.006. Epub 2019 Aug 20. PMID 31442616